CLINICAL TRIAL: NCT02839109
Title: PET-CT and DWI-MRI in Evaluating and Predicting Response to Neo-adjuvant Chemoradiotherapy in Esophageal Cancer Patients
Brief Title: PET-CT vs DWI-MRI in Response Evaluation in Esophageal Cancer
Acronym: PET/MRI-EC
Status: Completed | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Other Study IDs: NL49621.042.14
Record Dates: First submitted 2016-05-02; First posted 2016-07-20 (Estimated); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Esophageal Tumor
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
In patients with esophageal cancer (EC) neo-adjuvant chemoradiation (nCRT) followed by surgery with curative intent leads to objective responses in 45 to 60%, whereas 20-35% of the patients had no residual tumor (ypT0N0) at pathologic examination. The absolute survival benefit of response to nCRT is 15%, but still 14% of the patients develop locoregional failure in the CROSS trial. 18F-fluorodeoxyglucose positron emission tomography with computed tomography ((FDG-PET-CT) is able to distinct responders from non-responders, but still misses significant clinical evidence. Whole-body diffusion-weighted imaging (DWI) magnetic resonance imaging (MRI) has shown potential benefits, which might be enhanced by combining both methods. PET/CT and DWI-MRI more precisely correlate anatomic and metabolic FDG-avid lesions and seem to assess post-treatment changes, especially regarding nodal staging. Both techniques claim an important role in selection of patients with clinical complete response (cCR) and indirectly with pathologic complete response (pCR) after nCRT. However, the exact role and complementary effects of both techniques is still unknown.

For appropriate judgment of response, secure standard endoscopic ultrasonography (EUS) with fine needle aspiration (FNA) / biopsy of potential suspected lesions, both nodal or residual tumor, seen on PET/CT or DWI/MRI or during EUS will be performed <2 weeks before surgery, approximately 6-10 weeks after nCRT and compared with the situation at primary staging. Patients with clinical complete response (cCR) resembling pathologic response (pCR= ypT0N0) after nCRT may refrain from surgical resection and related morbidity and mortality. However, patients without early (2wk after commencement) response during nCRT course may not benefit from nCRT.

DWI-MRI seems effective in pre-treatment prediction of treatment outcome. Apparent diffusion coefficient (ADC), which indirectly measures tissue density, can be used to determine the likelihood of tumor response to treatment. High ADC before treatment has shown to predict an unfavorable response. Tumors with low ADC values on presentation generally respond better to treatment. An increased ADC in patients during and after nCRT could be used to predict early pathologic response i.e. discrimination of "responders and non-responders" to nCRT.

DETAILED DESCRIPTION:
DWI-MRI seems effective in pre-treatment prediction of treatment outcome. Tumor hypoxia mediates chemoradiation resistance, leading to selection of aggressive tumor cell clones with the capacity to evade tumor microenvironment by increased anaerobic glycolysis and angiogenesis. Apparent diffusion coefficient (ADC), which indirectly measures tissue density, can be used to determine the likelihood of tumor response to treatment. High ADC before treatment has shown to predict an unfavorable response. Tumors with low ADC values on presentation generally respond better to treatment. An increased ADC in patients during and after nCRT could be used to predict early pathologic response i.e. discrimination of "responders and non-responders" to nCRT.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically proven esophageal cancer (SCC and AC).
2. Age of 18 years or older.
3. Able to give written informed consent before registration.
4. T2-T4aN0M0 or T1-T4aN1-3M0 esophageal cancer.
5. Potentially curatively (R0) resectable tumor.
6. Tumor have sufficient FDG-baseline uptake.
7. Able to tolerate PET-CT and DWI-MRI as required by protocol.
8. Eligible for neo-adjuvant chemoradiotherapy (nCRT), including KPScore ≥ 70% / WHO>2; adequate renal, hepatic, hematological function.
9. No prior chemotherapy or mediastinal radiotherapy allowed.

Exclusion Criteria:

1. Non-resectable tumors: clinical or pathologic (T4b/R1-2 resections).
2. Proven distant metastases.
3. Prior malignancy except in-situ cervical lesions or non-melanoma skin cancer in the past 5 years.
4. Poorly controlled diabetes
5. Medical comorbidity preventing from surgery/preop CRT
6. General contraindications to MRI:

   * implanted pacemaker/serious claustrophobia
   * aneurysmal clips/metal implants in field of view

6. Major obesity (BMI > 40). 7. Active esophagitis. 8. Breast feeding/Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study group consists of patients with potentially curative (R0) resectable EC (T2-T4aN0M0/T1-T4aN1-3M0). These patients should be eligible for neo-adjuvant chemo-radiotherapy (CRT) including; performance/WHO ≤ 2; age > 18 yrs; hematology, electrolytes, liver and renal tests within normal range; no prior radio- or chemotherapy that would influence treatment for EC; no other malignancies (except basal cell carcinoma of the skin and carcinoma in situ), no active infect at the time of imaging, written informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2015-02; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Tumor response | Assessing clinical and pathologic response
  Within 2 weeks (early response) and at 6-10 weeks (late response)

SECONDARY OUTCOMES:
Disease free survival (DFS) | at 6 months, 1 year and 2 years

CONTACTS AND LOCATIONS:
Overall Officials: John Plukker, MD, PhD, Principal Investigator — Department of Surgical Oncology, University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
The results based on data of this study will be published in medical scientific papers. Moreover the data may be used for meta-analyses or conjoined research.